CLINICAL TRIAL: NCT00496301
Title: Phase II Clinical Trial, Non-Randomized, Multicentre, on the Combination of Gemcitabine, Capecitabine and Sorafenib (Bay 43-9006) in Treatment of Patients With Unresectable and/or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Clinical Trial on the Mixture of G, C and S in Treatment of Patients With RCC
Acronym: SOGUG-02-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Dr. Bellmunt Molins, Spanish Oncology Genito-Urinary Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-02-06
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal; sorafenib; Unresectable and/or metastatic renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Gemcitabine; Capecitabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine, Capecitabine and Sorafenib (6 cycles) — Gemcitabine: 1000 mg/m2 i.v. days 1 and 8. Capecitabine: 650 mg/m2 i.v. day 1 to 14. (change to 500mg/m2 after amendment nº2 (dated on 10/10/2007) Sorafenib:400 mg/12h v.o. day 1 to 21
  Other Names: Gemzar; Xeloda; Nexavar

SUMMARY:
Main Objective:

To evaluate progression-free survival in patients with unresectable renal cell carcinoma (RCC) treated with a combination of gemcitabine, capecitabine, and sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give their written informed consent before any procedure related to the study is performed; therefore, it must be given at the selection visit. The patient must be informed that he has the right to withdraw from the study at any time, without any kind of prejudice.
* Patients with renal clear cell carcinoma (RCC), unresectable and/or metastatic, histologically or cytologically documented (excluding the less common subtypes).
* Patients must not be candidates for any immunotherapeutic treatment, according to the response predictive factors, or must be intolerant to immunotherapeutic treatment.
* Patients classified as having median or low risk, according to Motzer's scoring.
* Patients (men or women) with ages equal or superior to 18 years old.
* ECOG ≤ 1.
* Assessable or measurable disease.
* Patients with adequate haematological function, defined as:

  * Neutrophils ≥ 1.5 x 10^9/L
  * Blood platelets ≥ 100 x 10^9/L
  * Haemoglobin ≥ 10 g/dl
* Patients with adequate hepatic, renal, medullar and coagulation function, according to the following criteria:

  * Total bilirubin < 1.5 times the superior limit of normality
  * ALT and AST < 2.5 times the superior limit of normality (< 5 times the superior limit of normality in case of liver failure due to cancer)
  * Amylase and lipase < 1.5 times the superior limit of normality
  * Serum creatinine < 2 times the superior limit of normality
  * TP or INR and TTP < 1.5 times the superior limit of normality. If patient is receiving anticoagulants, strict monitoring will be carried out, with evaluations on a weekly basis, at least, until the INR is stable, referring to a determination previous to dose administration, according to local standard care.
* Patients with a life expectancy superior to 12 weeks, at least.
* Patients may have received radiotherapy; however, this must not be the only target lesion.
* Patients from both sexes must use adequate contraceptive methods (oral or injectable contraceptives, intrauterine device, condom, sterilization) whilst participating in the protocol. After the retreat of treatment with BAY 43-9006, the contraceptive methods must be used for 4 weeks in women and for 3 months in men.
* Patients who are capable of accomplishing the study's requirements and without any impediments to follow the instructions while on study

Exclusion Criteria:

* Patients who do not give their written informed consent to participate in the study.
* Patients with less common RCC subtypes, such as pure papillary cell tumours, Bellini carcinoma, medullary carcinoma or the oncocytic chromophobes and sarcomatoid variants, will be excluded from the study.
* Patients that have received previous treatment with chemotherapy or that had tumours that evolved during or after immunotherapy treatment.
* Patients that, due to their characteristics, may obtain a potential benefit from immunotherapy treatment.
* Patients that have received previous anti-angiogenic treatment.
* High-risk patients according to Motzer's classification.
* Concomitant treatment with another chemotherapy or immunotherapy.
* Arterial uncontrolled hypertension, which is defined as a systolic arterial pressure value > 150 mmHg or diastolic arterial pressure value > 90 mmHg, despite adequate medical treatment.
* Patients with a primary cancer diagnosis different from RCC, except in situ cervical carcinoma, baseline cellular carcinomas or superficial bladder tumours, prostate cancer pT1 gleason < 6 or other malign tumours which have received curative treatment > 5 years previous to the inclusion in this study.
* Cardiac arrhythmia antecedents, that require treatment with anti-arrhythmics (except for beta-blockers or digoxin), symptomatic coronary disease or ischemia (myocardial infarction in the previous 6 months) or congestive cardiac insufficiency > New York Heart Association (NYHA) class II
* Patients with active bacterial or fungal infectious processes, which are considered severe from the clinical point of view (≥ Common Terminology Criteria from the National Cancer Institute [CTC from NCI] grade 2, version 3)
* Patients that present previously known positive serology for HIV or chronic hepatitis B or C.
* Antecedents of organ allograft.
* Meningeal carcinomatosis or symptomatic uncontrolled cerebral disease.
* Patients with epileptic disorders that require medication (such as antiepileptics).
* All unstable conditions that could put the patient's security and/or his study accomplishment in danger.
* Abuse of substances, clinical conditions, psychological or social, that may interfere with the patient's participation in the study or with the evaluation of the study's results.
* Patients that present any contraindication or allergy to the study's investigational product.
* Patients that are participating or that have participated in any clinical trial in the 4 weeks previous to inclusion.
* Pregnant or breastfeeding women. Women of fertile age must have a negative result in the pregnancy test performed 7 days before the beginning of the administration of the study medication. Both men and women included in the study must use an adequate contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 3 cycles and every two months in patients with "sorafenib" administered as monotherapy

SECONDARY OUTCOMES:
security profile | every 3 cycles and every two months in patients with "sorafenib" administered as monotherapy
Objective response index (CR/PR) and tumor growth control (CR/PR/SD) | every three cycles and every two months in patients with "Sorafenib" treated as single agent
Duration of response | every three cycles and every two months in patients with "Sorafenib" treated as single agent
Global survival | At last contact date or death date
Time to progression | every three cycles and every two months in patients with "Sorafenib" treated as single agent

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt Molins, MD, Study Chair — SOGUG
Locations (10):
- Spain (10):
  - Hospital Santiago de Compostela, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Josep Trueta, Girona
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Virgen Macarena, Seville
  - Hospital Xeral Cies, Vigo

REFERENCES:
- [Derived] Bellmunt J, Trigo JM, Calvo E, Carles J, Perez-Gracia JL, Rubio J, Virizuela JA, Lopez R, Lazaro M, Albanell J. Activity of a multitargeted chemo-switch regimen (sorafenib, gemcitabine, and metronomic capecitabine) in metastatic renal-cell carcinoma: a phase 2 study (SOGUG-02-06). Lancet Oncol. 2010 Apr;11(4):350-7. doi: 10.1016/S1470-2045(09)70383-3. Epub 2010 Feb 15. PMID 20163987